CLINICAL TRIAL: NCT06721104
Title: 'Evaluation of Temporomandibular Joint Dysfunction, Balance, Cervical Posture, Dual Task, and Social Adjustment in Individuals With Autism Spectrum Disorder'
Brief Title: Balance, TMJ, Social Adaptive Assessment in Individuals With Autism Spectrum Disorder
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Simay Tepik, Principal Investigator, Kırıkkale University
Other Study IDs: S1
Record Dates: First submitted 2024-11-25; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Temporomandibular Joint Disorders; Postural; Defect
MeSH Terms: conditions — Autism Spectrum Disorder; Temporomandibular Joint Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder
  Interventions: Other: Dual Task; Other: Functional Balance; Other: Social Adaptation Assessment; Other: Cervical Posture Assessment:; Other: Temporomandibular Joint (TMJ) Assessment
- Healthy Children
  Interventions: Other: Dual Task; Other: Functional Balance; Other: Social Adaptation Assessment; Other: Cervical Posture Assessment:; Other: Temporomandibular Joint (TMJ) Assessment

INTERVENTIONS:
Other: Dual Task — The dual-task abilities of individuals will be assessed by adding motor and cognitive tasks to the 10-Meter Walk Test. The tasks given to participants are as follows:
  Single Motor Task (comfortable walking): The individual is asked to walk at a normal pace, and the time is recorded.
  Motor-Motor Dual Task: The individual carries a half-filled water bottle in each hand while walking, and the time is recorded.
  Motor-Cognitive Dual Task (mental): The individual counts backward from 10 in increments of one while walking, and the time is recorded.
  Motor-Cognitive Dual Task (memory): The individual is asked to recall three previously mentioned words while walking, and the time is recorded.
Other: Functional Balance — Functional balance will be assessed using the Timed Up and Go (TUG) test. The TUG test measures the time it takes for an individual to stand up from a chair upon the "ready, go" signal, walk a distance of 3 meters, turn around, walk back to the chair, and sit down again. The TUG test is a reliable and sensitive measure of balance and functional mobility in children.
  At the beginning of the test, participants will be seated on an armless chair with their hips and knees flexed at approximately 90 degrees and their feet flat on the ground. The children will be instructed to stand up from the chair, walk as quickly as possible, touch a target on the wall, walk back, and sit down again.
Other: Social Adaptation Assessment — Adaptive behavior will be evaluated using the Vineland Adaptive Behavior Scales. This is a parent interview designed to assess functionality in daily life. Specifically, adaptive behavior is evaluated in four domains: Communication, Daily Living Skills, Socialization, and Motor Skills. The Vineland scales are known for their reliability and up-to-date validity. They have been reported to be sensitive to the challenges faced by children with Autism Spectrum Disorder (ASD).
Other: Cervical Posture Assessment: — Cervical posture will be evaluated using the Android-based PostureScreen Mobile application (version 8.5, developed by Posture Co. Inc., USA). This application assesses the static posture of individuals. After determining reference points, the application draws reference lines and records postural deviations. At least two photos of each participant will be taken for the assessment. Participants should not wear clothing items that cover the neck (e.g., scarves, shawls).
  While the primary focus of the application is to assess postural deviations, it also includes a dental evaluation feature. The validity and reliability of the application have been established in previous studies. In addition to using the application, the posture of individuals will also be evaluated through observational analysis, and the findings will be documented.
Other: Temporomandibular Joint (TMJ) Assessment — The TMJ will be evaluated using the Helkimo Clinical Craniomandibular Index. This index consists of five subcategories: pain during muscle palpation, pain during TMJ palpation, pain during mandibular functions, TMJ functions (sounds, gliding during maximum opening, dislocation and/or locking), and the mandibular range of motion. Each subcategory is scored as 0, 1, or 5, resulting in a total score ranging from 0 to 25.
  As this index is based on performance measurements, there is no Turkish validity and reliability study for it. However, a prevalence study using this index was conducted in Turkey by Üner et al. to evaluate its applicability within the Turkish population.

SUMMARY:
The aim of our study is to evaluate temporomandibular joint (TMJ), cervical posture, balance, dual-task performance, and social adaptation skills in individuals with autism. The study will be conducted at Bartın Lider Special Education and Rehabilitation Center following the approval of the ethics committee. Individuals determined by the sample size calculated through power analysis will be included in the study. First, the socio-demographic characteristics (age, height, body weight, body mass index, education level, exercise and smoking habits, etc.) of the participants who voluntarily join the study will be recorded. Participants will be divided into two groups: individuals with typical motor development and those with autism spectrum disorder (ASD), and the same assessment tools will be used for both groups. Individuals with typical motor development will serve as the control group.

The assessment tools include the Timed Up and Go (TUG) test, the 10-Meter Walk Test, the Vineland Adaptive Behavior Scale, the PostureScreen Android-based posture assessment application, and the Helkimo Clinical Dysfunction Index for craniomandibular disorders. Based on the evaluation results, the relationships between TMJ, cervical posture, functional balance, dual-task performance, and social adaptation skills in individuals with autism will be analyzed and compared with those of individuals with typical motor development.

DETAILED DESCRIPTION:
It has been stated in the literature that individuals with autism spectrum disorder have postural control deficiency, but there is no study examining the dual task skills of these individuals and the contribution of these skills to social life.

It has been stated in the literature that bruxism can cause TMJ in individuals with normal development, and there are studies related to TMJ's cervical problems and balance. However, there are no studies explaining the relationship between teeth grinding and dental problems in individuals with ASD, temporomandibular joint problems and cervical posture and balance.

Studies suggest that multi-faceted evaluations be made in individuals with ASD. The aim of our study is to evaluate TMJ dysfunction, cervical posture, functional balance, dual task and social adaptation skills in individuals with ASD. In terms of these evaluations, our study has the feature of a pilot study in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Autism Spectrum Disorder (ASD) confirmed by a physician.
* Currently enrolled in a special education and rehabilitation center.
* No vision problems.
* Ability to understand and follow instructions.
* No cognitive impairments.
* No walking difficulties.

Exclusion Criteria:

* Individuals with comorbid secondary health conditions.
* Individuals who have undergone surgery in the past six months.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The assessments will be conducted at the Physical Therapy Unit of the Lider Special Education and Rehabilitation Center, where voluntary families will be contacted and evaluations will be carried out within the rehabilitation center.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Cervical Posture Assessment | At enrollment
  Android-based PostureScreen Mobile (version 8.5, developed by Posture CO.inc. USA) application will be used for cervical posture assessment. The application evaluates the static posture of individuals

SECONDARY OUTCOMES:
Temporomandibular Joint (TMJ) Assessment: | At enrollment
  Helkimo Clinical Craniomandibular Index will be used for TMJ evaluation. This index consists of 5 subsections: pain on muscle palpation, pain on TMJ palpation, pain in mandibular functions, TMJ functions (sound, gliding at maximum extension, luxation and/or locking) and the capacity of mandibular movement.
Social Adaptation Assessment: | At enrollment
  Adaptive behavior will be assessed with the Vineland Adaptive Behavior Scales. It is a parent interview designed to assess functioning in daily life.
Functional Balance | At enrollment
  It will be assessed with the TUG test. The TUG ready measures the time it takes for an individual to get up from a chair, walk a distance of 3 meters, turn around, walk back to the chair and sit down again after the start signal.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Sertel, Dr., Study Chair — Kırıkkale University
Locations (1):
- Kırıkkale Universty, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes